CLINICAL TRIAL: NCT01789879
Title: A Pharmacokinetic Evaluation of Levonorgestrel Implant and Non-nucleoside Reverse Transcriptase Inhibitor (NNRTI)-Based Antiretroviral Therapy in HIV-infected Ugandan Women
Brief Title: A Pharmacokinetic Evaluation of Levonorgestrel Implant and Antiretroviral Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Makerere University (Other); University of Liverpool (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0022-14-EP; 1R21HD074462-01 (NIH)
Record Dates: First submitted 2013-02-07; First posted 2013-02-12 (Estimated); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: HIV; Contraception
Keywords: Levonorgestrel; Efavirenz; Nevirapine; Pharmacokinetics
MeSH Terms: interventions — Levonorgestrel; Nevirapine; efavirenz; Efavirenz, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control group (no current ART) (Active Comparator): Levonorgestrel subdermal implant in subjects not yet receiving ART (control group)
  Interventions: Drug: Levonorgestrel
- NVP-based ART group (Active Comparator): Levonorgestrel subdermal implant in subjects receiving nevirapine-based ART
  Interventions: Drug: Levonorgestrel; Drug: Nevirapine
- EFV-based ART group (Active Comparator): Levonorgestrel subdermal implant in subjects receiving efavirenz-based ART
  Interventions: Drug: Levonorgestrel; Drug: Efavirenz

INTERVENTIONS:
Drug: Levonorgestrel — Levonorgestrel 2-rod subdermal implant (75mg/rod) placed on study day 0 after baseline evaluations and remains in place until the subject requests removal or for the duration of drug activity (currently approved for 5 years).
  Other Names: Jadelle; SinoImplant
Drug: Nevirapine — Nevirapine 200mg twice daily as part of a complete antiretroviral therapy regimen. Subjects will be on this therapy prior to entry in this study.
  Other Names: Viramune; NVP
  Arms: NVP-based ART group
Drug: Efavirenz — Efavirenz 600mg once daily as part of a complete antiretroviral therapy regimen. Subjects will be on this therapy prior to entry in this study.
  Other Names: Sustiva; Atripla; Stocrin; EFV
  Arms: EFV-based ART group

SUMMARY:
The use of hormone contraception poses a significant challenge for the estimated 16 million HIV-infected women of childbearing age. This is due to known drug interactions with antiretroviral therapy (medicines used to treat HIV) that may jeopardize contraception effectiveness. By evaluating the impact of antiretroviral therapy on a levonorgestrel subdermal implant, the most widely available hormone implant in low and middle-income countries, this study will translate its findings into an evidence-based approach to co-manage these important medications. The investigators hypothesize that women receiving nevirapine or efavirenz-based antiretroviral therapy will have a significant decrease in the mean levonorgestrel plasma concentration measured six months after the implant's insertion as compared to those women who are not taking antiretroviral therapy. Although the implant's efficacy may be retained initially, the investigators propose that a decrease in levonorgestrel concentrations in women receiving antiretroviral therapy may jeopardize the implant's effectiveness near the end of its intended duration of use (5 years).

DETAILED DESCRIPTION:
Family planning services, including hormone contraceptives, are critical for HIV-infected women, in whom prevention of unintended pregnancy not only decreases maternal and child mortality, but also reduces the risk of mother-to-child HIV transmission. Similarly, antiretroviral therapy (ART) is a lifesaving intervention that improves the health and economic status of HIV-infected women throughout the world. Therefore, it is of significant public health importance to guide the appropriate use these essential medications. To this end, millions of HIV-infected women in low and middle income countries (LMIC) currently use or are gaining access to subdermal progestin-containing implants as a preferred method of long-acting reversible contraception. These implants are often combined with ART despite the lack of critically needed pharmacokinetic (PK) drug-interaction data to inform their safe and effective concomitant use. Highlighting this concern are several case reports of unintended pregnancy that occurred in patients with subdermal progestin-containing implants concurrently receiving non-nucleoside reverse transcriptase inhibitor (NNRTI)-based ART, the most commonly used ART in LMICs. While NNRTIs are known to significantly decrease oral pill progestin concentrations, no data are available to inform healthcare providers of the impact of NNRTIs on progestin concentrations following release from subdermal implants. To fill this critical gap in knowledge, the overall aim of this proposal is to conduct a PK study to evaluate the combination of a levonorgestrel (LNG) implant and NNRTI (nevirapine or efavirenz)-based ART in HIV-infected Ugandan women. The investigators propose that lower LNG concentrations will be observed in patients on NNRTI-based ART and although the implant's efficacy may be retained initially, this negative interaction will jeopardize implant effectiveness near the end of its intended duration of use (5 years). The specific aims of this project are (1) to characterize the PK of LNG released from a subdermal implant over one year in HIV-infected women with and without NNRTI-based ART and (2) to evaluate the potential for a bidirectional drug-interaction resulting from the long-term impact of chronic progestin exposure on antiretroviral concentrations. To achieve these aims, this study will enroll 20 HIV-infected women into each of three study groups: a control group not receiving ART and two treatment arms consisting of patients receiving nevirapine- or efavirenz- based ART. Using sparse PK sampling strategies, LNG, nevirapine or efavirenz concentrations will be measured over one-year and compared between and within groups, as appropriate. The LNG data will also be used to develop a PK model that will predict LNG disposition over the following three years of intended use, allowing for identification of the safe duration of LNG implant use in women on NNRTI-based ART. At the conclusion of this project, the first evidence-based medical knowledge will be available to guide the safe and effective concomitant use of subdermal LNG implants and NNRTIs, thereby improving management of reproductive health in millions of HIV-infected women worldwide.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of a personally signed and dated informed consent document indicating that the subject (or a legal representative) has been informed of all pertinent aspects of the study.
* Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
* Women age 18 years or older
* Diagnosed with HIV-1 infection
* Desiring LNG subdermal implant as a contraceptive method
* Subjects not yet eligible for ART (based on the Ugandan Treatment Guidelines); or subjects receiving nevirapine or efavirenz-based ART for a minimum of 1 month prior to screening

Exclusion Criteria:

* For patients currently on ART: HIV-1 RNA > 400 copies/mL at screening visit
* Serum hemoglobin < 9.0 g/dl
* Elevations in serum levels of alanine transaminase (ALT) above 5 times the upper limit of normal
* Elevations in serum creatinine above 2.5 times the upper limit of normal
* Use of drugs known to be contraindicated with levonorgestrel, nevirapine (NVP group only), or efavirenz (EFV group only) within 30 days of study entry. Due to the dynamic nature of drug interactions related to antiretroviral therapy, the study team will review all concomitant medications at screening based on the US Department of Health and Human Services drug interaction tables or the AIDS Clinical Trials Group Drug Interactions Database.
* Currently pregnant or postpartum <30 days at study entry
* No concurrent use of other hormonal contraception is allowed during the study period

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-03-04 (Actual); Primary Completion 2014-09-01 (Actual); Study Completion 2015-03-04 (Actual)

PRIMARY OUTCOMES:
Levonorgestrel plasma concentrations | 6 months and 1 year after implant
  Levonorgestrel plasma concentrations

SECONDARY OUTCOMES:
Non-nucleoside reverse transcriptase inhibitor (NNRTI) plasma concentrations | Over 1 year (baseline, Months 1, 3, 6, 9, and 12)
  Applies to subjects being treated with either efavirenz- or nevirapine-based antiretroviral therapy

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly K Scarsi, PharmD, MSc, Principal Investigator — University of Nebraska
Locations (1):
- Infectious Diseases Institute, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Scarsi KK*, Darin KM, Nakalema S, Back D, Byakika-Kibwika P, Else L, Dilly-Penchala S, Cohn S, Merry C, Lamorde M. Levonorgestrel implant + EFV-based ART: Unintended pregnancies and associated PK Data. Conference on Retroviruses and Opportunistic Infections. Seattle, WA. February 23-26, 2015. Abstract #85LB.
- [Result] Scarsi K, Lamorde M, Darin K, Penchala SD, Else L, Nakalema S, Byakika-Kibwika P, Khoo S, Cohn S, Merry C, Back D. Efavirenz- but not nevirapine-based antiretroviral therapy decreases exposure to the levonorgestrel released from a sub-dermal contraceptive implant. J Int AIDS Soc. 2014 Nov 2;17(4 Suppl 3):19484. doi: 10.7448/IAS.17.4.19484. eCollection 2014. PMID 25393993
- [Result] Scarsi KK, Darin KM, Nakalema S, Back DJ, Byakika-Kibwika P, Else LJ, Dilly Penchala S, Buzibye A, Cohn SE, Merry C, Lamorde M. Unintended Pregnancies Observed With Combined Use of the Levonorgestrel Contraceptive Implant and Efavirenz-based Antiretroviral Therapy: A Three-Arm Pharmacokinetic Evaluation Over 48 Weeks. Clin Infect Dis. 2016 Mar 15;62(6):675-682. doi: 10.1093/cid/civ1001. Epub 2015 Dec 8. PMID 26646680